CLINICAL TRIAL: NCT05648292
Title: The Relationships Between Personal Identity, Autobiographical Memory and Future Thinking in People With Multiple Sclerosis
Acronym: SELFSEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: University Paris 8 Vincennes Saint Denis (Other); ARSEP foundation (Unknown)
Responsible Party: Principal Investigator, Alexandra Ernst, Associate Professor, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: 2022-A00495-38
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Healthy Controls
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical group: 45 individuals with relapsing-remitting multiple sclerosis
  Interventions: Behavioral: Neuropsychological tests and psychological questionnaires
- Control group: 45 individuals with no chronic disease, matched in age, gender and level of education
  Interventions: Behavioral: Neuropsychological tests and psychological questionnaires

INTERVENTIONS:
Behavioral: Neuropsychological tests and psychological questionnaires — * The clinical group will complete:
    * the BCcogSEP: a comprehensive neuropsychological examination
    * the IAM and I WILL BE tasks; experimental neuropsychological tasks to assess autobiographical memory, future thinking and personal identity
    * A series of questionnaires including the BRIEF COPE, the Connor Davidson Resilience Scale, the Satisfaction with Life Scale and the Hospital Anxiety and Depression Scale, which respectively assess coping strategies, resilience, life satisfaction and anxiety/depression
  * The control group will complete:
    * the IAM and I WILL BE tasks; experimental neuropsychological tasks to assess autobiographical memory, future thinking and personal identity
    * A series of questionnaires including the BRIEF COPE, the Connor Davidson Resilience Scale, the Satisfaction with Life Scale and the Hospital Anxiety and Depression Scale, which respectively assess coping strategies, resilience, life satisfaction and anxiety/depression

SUMMARY:
Personal identity is composed of multiple facets of the self that are constructed and nourished through memories of past experiences (i.e., autobiographical memory) and the imagination of events that may occur in the future (i.e., future thinking) .

While our previous work has shown that people with relapsing-remitting multiple sclerosis (pwRRMS) have autobiographical memory and future thought disorders, their impact on personal identity has not yet been explored. Based on a cognitive and clinical neuropsychology approach, this research project aims to better understand the cognitive mechanisms involved in the relationship between identity, autobiographical memory and future thinking in pwRRMS. We will examine the extent to which pwRRMS manage to maintain and reshape their identity through life experiences, with a particular interest in the potential integration of the disease as a facet of their identity. In addition, we will explore the positive and/or negative consequences of disease-related identity changes on emotional well-being and quality of life, as well as their links with the duration and severity of the disease. Overall, this research project will contribute to identify new therapeutic levers that can be used for the development of adapted and personalized care.

ELIGIBILITY:
For the clinical group:

Inclusion Criteria:

* Diagnosis of relapsing-remitting MS according to the McDonald's revised diagnostic criteria
* People aged between 18 and 55
* French native speaker
* Access to a computer or tablet, equipped with internet access, a camera and a microphone

Non-inclusion Criteria:

* MS relapse in the month prior to the inclusion
* Treatment with corticosteroids during the month preceding the inclusion
* Form of MS other than the relapsing-remitting form
* Neurological history (other than MS for patients), history or current presence of psychiatric disorders (e.g., depression, anxiety disorders, schizophrenia), substance abuse (e.g., alcohol, cannabis; past or present)
* Other diagnosed chronic pathology(ies) (other than MS for patients)
* Severe cognitive impairment
* Persons mentioned in Articles L1121-6 to L1121-8 in the French law (minors, persons deprived of liberty, adults subject to protective measures)

For the control group:

Inclusion Criteria:

* People aged between 18 and 55
* Matched in age, gender and level in education
* French native speaker
* Access to a computer or tablet, equipped with internet access, a camera and a microphone

Non-inclusion Criteria:

* Neurological history (other than MS for patients), history or current presence of psychiatric disorders (e.g., depression, anxiety disorders, schizophrenia), substance abuse (e.g., alcohol, cannabis; past or present)
* Other diagnosed chronic pathology(ies) (other than MS for patients)
* Severe cognitive impairment
* Persons mentioned in Articles L1121-6 to L1121-8 in the French law (minors, persons deprived of liberty, adults subject to protective measures)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-12-07 (Estimated); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
Relationships between personal identity, autobiographical memory and future thinking | 15 days
  Scores obtained at the I AM and I WILL BE tasks assessing the access, qualitative properties of self-concepts, episodic richness and temporal organization of past and future events around self-concepts (between-group comparisons, pwRRMS versus control group)

SECONDARY OUTCOMES:
Relationships between personal identity, psychological functioning and clinical characteristics | 15 days
  Correlations between IAM and I WILL BE scores and scores obtained at the different questionnaires (BRIEF COPE, Connor Davidson Resilience Scale, Satisfaction with Life Scale, Hospital Anxiety and Depression Scale) Correlations between IAM and I WILL BE scores and level of functional disability (Expanded Disability Status Scale) Correlations between IAM and I WILL BE scores and disease duration

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra ERNST, PhD, Principal Investigator — Laboratoire DysCo - Université Paris 8
Locations (1):
- Hopital Raymond Poincaré Garches, Garches, Hauts De Seine, France

IPD SHARING:
Plan to Share IPD: No